CLINICAL TRIAL: NCT02355717
Title: Role of Cardiometabolic Risk Factors in Childhood Bone Development (Healthy Heart 'N' Bones Study)
Brief Title: Role of Cardiometabolic Risk Factors in Childhood Bone Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Norman Pollock, Associate Professor, Department of Medicine, Augusta University
Other Study IDs: 616274
Record Dates: First submitted 2015-01-22; First posted 2015-02-04 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Cardiovascular Disease; Type 2 Diabetes; Osteoporosis
Keywords: children, bone; Simple obesity; cardiovascular disease; osteoporosis; diabetes
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Osteoporosis; Diabetes Mellitus | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prospective Cohort: 400 otherwise healthy children and adolescents aged 9-15 years will be recruited to participate in a 2-year longitudinal study.
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study

SUMMARY:
The proposed research brings together complementary expertise to systematically elucidate the longitudinal effects of (1) total and regional body fat and (2) the metabolic impairment that accompanies obesity on bone development during growth. The contribution of this research will be significant because it will provide a solid foundation for understanding the influence of fat (total and regional distribution) on overall bone strength, and whether insulin resistance, beta-cell dysfunction, abnormal lipids, and inflammation could be underpinning factors in the fat-bone strength relationship via effects on bone modeling activity. This knowledge will provide critical information needed to maximize potential therapeutic interventions to counter the linked risks of obesity and osteoporosis, both major public health concerns.

DETAILED DESCRIPTION:
The overall goal of this study is to clarify the relationship of adiposity with bone development during adolescence, and to explicate the mechanisms that regulate the effect of excess adiposity on bone. In this effort, we will conduct a 2-year longitudinal study in 400 children and adolescents aged 9-15 years. Using the peak adolescent growth period as a model for probing determinants of bone health may allow for a clearer picture of the processes that regulate bone development, as these processes are highly active at this growth stage. Unlike other studies with surrogates for adiposity, we plan to measure total and central adiposity directly, using dual energy X-ray absorptiometry (DXA) and magnetic resonance imaging. Both bone quantity and bone quality, the two principal determinants of bone strength, will be assessed by peripheral quantitative computed tomography (pQCT) at weight-bearing (tibia) and non-weight-bearing (radius) skeletal sites. Peripheral QCT provides 3-dimensional bone measurements that are not confounded by changes in bone size, a significant confounder of most past studies, which have relied on 2-dimensional bone imaging techniques. To identify mechanistic factors, which may explain the effect of adiposity on bone development, we will measure arterial stiffness, endothelial function, and fasting levels of glucose, insulin, lipids, and C-reactive protein (CRP) to assess how vascular dysfunction, insulin resistance, abnormal lipids, and inflammation are related to bone modeling activity, as measured by serum markers of bone formation and resorption. All measurements will be assessed at baseline and after 1 and 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy children and adolescents between 9 and 15 years old
2. Subject and parent/guardian understands the study protocol and agrees to comply with it
3. Informed Consent Form signed by the parent/guardian and assent signed by the subject

Exclusion Criteria:

1. Subjects with (a history of) metabolic or gastrointestinal diseases including hepatic disorders
2. Subjects presenting chronic degenerative and/or inflammatory diseases
3. Subjects receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters (salicylates, antibiotics)
4. Subjects receiving corticosteroid treatment
5. Subjects using oral anticoagulants
6. Subjects who have participated in a clinical study more recently than one month before the current study

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 400 children and adolescents aged 9 to 15 years
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-12; Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Bone mineral mass | Change from baseline bone mineral mass at 2 years
  Measurement of bone quantity assessed by peripheral quantitative computed tomography
Bone strength-strain index | Change from baseline bone strength-strain index at 2 years
  Measurement of bone quality assessed by peripheral quantitative computed tomography

SECONDARY OUTCOMES:
Serum N-terminal propeptide of type 1 procollagen (P1NP) | Change from baseline P1NP at 2 years
  Marker of bone formation as measured in serum
Serum C-terminal telopeptide of type 1 collagen (CTX) | Change from baseline CTX at 2 years
  Marker of bone resorption as measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: Norman K Pollock, Ph.D., Principal Investigator — Department of Medicine, Medical College of Georgia, Augusta University
Locations (1):
- Medical College of Georgia; Augusta University, Augusta, Georgia, United States

REFERENCES:
- [Background] Pollock NK, Laing EM, Baile CA, Hamrick MW, Hall DB, Lewis RD. Is adiposity advantageous for bone strength? A peripheral quantitative computed tomography study in late adolescent females. Am J Clin Nutr. 2007 Nov;86(5):1530-8. doi: 10.1093/ajcn/86.5.1530. PMID 17991669
- [Background] Pollock NK, Bernard PJ, Wenger K, Misra S, Gower BA, Allison JD, Zhu H, Davis CL. Lower bone mass in prepubertal overweight children with prediabetes. J Bone Miner Res. 2010 Dec;25(12):2760-9. doi: 10.1002/jbmr.184. Epub 2010 Jul 16. PMID 20641032
- [Background] Pollock NK, Laing EM, Hamrick MW, Baile CA, Hall DB, Lewis RD. Bone and fat relationships in postadolescent black females: a pQCT study. Osteoporos Int. 2011 Feb;22(2):655-65. doi: 10.1007/s00198-010-1266-6. Epub 2010 May 7. PMID 20449571
- [Background] Pollock NK, Bernard PJ, Gutin B, Davis CL, Zhu H, Dong Y. Adolescent obesity, bone mass, and cardiometabolic risk factors. J Pediatr. 2011 May;158(5):727-34. doi: 10.1016/j.jpeds.2010.11.052. Epub 2011 Jan 13. PMID 21232765
- [Background] Pollock NK, Laing EM, Taylor RG, Baile CA, Hamrick MW, Hall DB, Lewis RD. Comparisons of trabecular and cortical bone in late adolescent black and white females. J Bone Miner Metab. 2011 Jan;29(1):44-53. doi: 10.1007/s00774-010-0186-z. Epub 2010 May 11. PMID 20458605
- [Background] Pollock NK, Bernard PJ, Gower BA, Gundberg CM, Wenger K, Misra S, Bassali RW, Davis CL. Lower uncarboxylated osteocalcin concentrations in children with prediabetes is associated with beta-cell function. J Clin Endocrinol Metab. 2011 Jul;96(7):E1092-9. doi: 10.1210/jc.2010-2731. Epub 2011 Apr 20. PMID 21508147
- [Background] Laing EM, Tripp RA, Pollock NK, Baile CA, Della-Fera MA, Rayalam S, Tompkins SM, Keys DA, Lewis RD. Adenovirus 36, adiposity, and bone strength in late-adolescent females. J Bone Miner Res. 2013 Mar;28(3):489-96. doi: 10.1002/jbmr.1776. PMID 23296755
- See also: Faculty Directory Profile — https://www.augusta.edu/faculty/directory/view.php?id=NPOLLOCK